CLINICAL TRIAL: NCT01932424
Title: Comparison of Measured Versus Predicted Blood Propofol Concentrations During Total Intravenous Anaesthesia in Children Undergoing Spinal Surgery
Brief Title: Blood Propofol Concentrations in Children During Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: 12AR04
Record Dates: First submitted 2013-08-13; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Spine Deformities; Idiopathic Scoliosis; Neuromuscular Dystrophy
Keywords: Children
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): The intervention in this study involves taking blood sample from an existing arterial line for measurement of blood propofol levels. The drug in evaluation is Propofol 2% (Diprivan 2%, Astra Zeneca UK) administered as a target controlled infusion using the commercially available paediatric TCI models (Paedfusor and Marsh models). The dose range is usually between a target concentration of 3-8 mcg/ml. However the anaesthetic management is not changed for the study. The blood concentrations of propofol will be measured using Pelorus 1500 (Sphere Medical, UK), a CE marked device. The anaesthetist will be blinded from the measurements, unless the measured value was outside the safe limit ( < 3 mcg/ml or > 10mcg/ml).
  Interventions: Device: Pelorus 1500; Drug: Propofol 2% (Diprivan 2%, Astra Zeneca UK)

INTERVENTIONS:
Device: Pelorus 1500 — a bedside blood propofol measurement device
  Other Names: Sphere Medical, UK
Drug: Propofol 2% (Diprivan 2%, Astra Zeneca UK)

SUMMARY:
During major spinal surgery evoked potential monitoring is performed to detect spinal cord damage. Intra-venous anaesthesia is the preferred anaesthetic technique because volatile anaesthetic agents supress the evoked potentials. Total Intra-Venous Anaesthesia (TIVA) with propofol is commonly administered as a Target Controlled Infusion (TCI). The TCI is an automated drug delivery system which administers propofol to achieve a desired blood concentration, based on an in built pharmaco-kinetic data (TCI model) derived from previous studies. The TCI model also provides a real time predicted blood concentration to facilitate the anaesthetist to adjust the target concentration of propofol.

The TCI algorithm is based on pharmaco-kinetic data derived from previous studies in a relatively small number of patients, by a "best fit" relationship between blood levels, infusion rates and other factors (such as age and weight). Several factors make it possible for a wide discrepancy between the predicted and the true blood concentrations. This difference can be higher in children compared to adults. Also blood loss and administration of large volumes of intravenous fluids can affect the blood concentrations. This study aims to identify the difference between the predicted and true blood concentrations by using Pelorus 1500, a bedside blood propofol measurement device, in children undergoing major spinal surgery under TIVA.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing major spinal surgery under propofol TCI
* Surgery expecting to last more than 3 hours.

Exclusion Criteria:

* Major hepatic or renal disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The absolute difference between the measured and predicted concentrations of propofol in micrograms per ml of blood. | Up to 5 hours during the maintenance phase of anaesthesia, to allow a maximum of 10 samples at 20 to 30 min intervals.

SECONDARY OUTCOMES:
Median Performance Error (MDPE) | Up to 5 hours during the maintenance phase of anaesthesia, to allow a maximum of 10 samples at 20 to 30 min intervals.
  The median value of ratio between the measured and predicted concentration of propofol to the predicted concentration (Performance error) in blood. Expressed as a percentage. This is a measure of overall bias of the target controlled infusion.
Median Absolute Performance Error (MDAPE) | Up to 5 hours during the maintenance phase of anaesthesia
  The median value of the ratio of the absolute difference (excluding the sign) between the measured and predicted concentrations to the predicted concentration (Absolute performance error) in blood. Expressed as percentage. This is a measure of the accuracy of the target controlled infusion.
Wobble | Up to 5 hours during the maintenance phase of anaesthesia
  The median value of the difference between the individual performance errors and the Median Performance Error (MDPE). This is a measure of the distribution of the performance errors around the median.
Divergence | Up to 5 hours during the maintenance phase of anaesthesia
  The median of the regression coefficient of the performance error against time. This is a measure of how the target controlled infusion performs with time.

CONTACTS AND LOCATIONS:
Overall Officials: Michael RJ Sury, FRCA PhD, Study Director — Great Ormond Street Hospital for Children NHS Foundation Trust; Selvakumar Panchatsharam, MBBS FRCA, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS trust, London, London, United Kingdom